CLINICAL TRIAL: NCT05595161
Title: Dissemination and Implementation of the Bright Bodies Intervention for Childhood Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000032608; 5R01HL151603-02 (NIH)
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Childhood
Keywords: Implementation science; Intensive lifestyle intervention; Pediatric obesity; Behavior modification; Body mass index
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Bright Bodies
  Interventions: Behavioral: Bright Bodies

INTERVENTIONS:
Behavioral: Bright Bodies — The Bright Bodies intensive, family-based lifestyle intervention uses group sessions including nutrition education, behavior modification, and exercise to improve weight and weight-related outcomes among children and adolescents with obesity.
  Other Names: SmartMoves TM (name of the curriculum used in the Bright Bodies intervention)

SUMMARY:
This study will evaluate the effectiveness of the Bright Bodies intervention in improving body mass index (BMI) among 7-13 year-old children with obesity simultaneously with the impact of the implementation strategy on adoption, reach, fidelity, cost, and maintenance of the intervention in three heterogenous settings serving patients disproportionately affected by obesity.

DETAILED DESCRIPTION:
The demonstrated efficacy of Bright Bodies in a well-designed randomized controlled trial (RCT) and a real-world effectiveness study reduce equipoise and challenge the ethics of a prospective RCT of implementing Bright Bodies in other settings. As such, this study is an observational, multiphase mixed methods design to evaluate effectiveness and implementation among three purposively selected heterogeneous sites serving low-income populations with racial and ethnic, rural-urban, and geographic diversity.

Children ages 7-13 years with BMI ≥85th percentile and their parent/caregivers hereafter referred to as parent will be recruited to participate in the evaluation study from among participants in the newly-established Bright Bodies programs at each of the three implementation sites. The aim is for each site to recruit approximately 40 children and their parents (a total of 120 children and 120 parents) to participate in the Bright Bodies program over the study's enrollment period. The primary outcome is change in BMI expressed as a percentage of the 95th percentile (%BMIp95) using EHR data collected as part of routine clinical care up to 36 months before and up to 15 months after enrollment in the intervention. Secondary outcomes include: (a) change in %BMIp95 at three and six months, (b) changes in parent BMI at three and six months, (d) parent-reported changes in health behaviors (sleep, physical activity, screen time, eating behaviors), via surveys at 3, 6 and 12 months, and (e) changes in parent-proxy reported weight-related quality of life, parent stress, and parent talk about weight via surveys at baseline, 6, and 12 months after enrollment. We will also describe implementation outcomes (reach, adoption, fidelity/adaptation, and cost) through qualitative and quantitative data collection from members of our study team throughout the process of implementation.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-13 years with BMI ≥85th percentile and their parents;
* Child-parent dyads enrolled in the Bright Bodies intervention at each site will be eligible for inclusion in the evaluation study.

Exclusion Criteria:

* Children and/or parents who do not speak the language in which the program will be delivered at each site;
* Children and/or parents who plan to move away from the area within the next 15 months;
* Children with a history of purging and/or dramatic weight loss prior to the trial;
* Children who are currently participating in another high-intensity lifestyle intervention or other similar research study, or are planning to have bariatric surgery within the next six months
* Children whose EHR data cannot be accessed by the study teams;
* Children with chronic medical conditions limiting their ability to take food by mouth (e.g., g-tube fed, total parenteral nutrition), participate in physical activity (e.g., wheelchair bound), or meaningfully participate in group sessions (e.g., cognitive impairment);
* Children with a sibling enrolled in the trial
* Children who join the Bright Bodies program after the 4th week of a session (not including orientation)

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Change in %BMIp95 | Up to 36 months prior to baseline through up to 15 months after enrollment
  Change in %BMIp95, calculated from height and weight. A negative percentage indicates that the participant's BMI has decreased since enrollment.

SECONDARY OUTCOMES:
Change in parent BMI | Baseline through 6 months after enrollment
  Change in BMI, calculated from height and weight measured as part of the Bright Bodies program. A negative change in parent BMI indicates that the parent's BMI has decreased since enrollment.
Change in weight-related quality of life | Baseline through 12 months after enrollment
  Sizing Them Up is a validated, parent-proxy reported instrument assessing weight-related quality of life for children aged 5-13 years. Possible score ranges from 1 (never) to 4 (always). Higher score indicates a higher quality of life.
Change in weight-related health behaviors. | Baseline through 12 months after enrollment
  Parent-proxy responses to the Bright Bodies Healthy Lifestyles Questionnaire about vegetable and fruit intake [scores range from 1 (none) to 4 (three or more); Higher score indicates healthier behavior]; sugar-sweetened beverage intake [scores range from 1 (none) to 4 (three or more); Lower score indicates healthy behavior]; intake of sweets/desserts [scores range from 1 (none) to 4 (seven or more); Lower score indicates healthy behavior]; physical activity [scores range from 1 (less than 30 minutes) to 4 (more than 2 hours); higher score indicates healthy behavior.]; screen time [scores range from 1 (more than 4 hours) to 4 (1 hour or less); higher score indicates healthy behavior.]; sleep [scores range from 1 (6 hours or less) to 3 (9 hours or more) for the amount a child sleeps each night and from 1 (no) to 2 (yes) for the question about a regular bedtime; Higher score indicates healthy behavior].
Change in binge eating behaviors. | Baseline through 12 months after enrollment
  Children's Brief Binge-Eating Questionnaire will be parent-proxy reported. Possible score ranges from 1 (definitely false) to 3 (definitely true). Higher scores indicate greater concern for binge eating behavior.
Change in parent conversations about weight. | Baseline through 12 months after enrollment
  Parent conversation about weight is measured with three questions using a parent self-report instrument from the New Moves, a school-based intervention designed to prevent obesity and other weight-related problems. Possible scores range from 1 (never) to 5 (very often). Lower score indicates less weight talk.
Per patient cost for participation in Bright Bodies | From enrollment through 12 months after enrollment
  Calculated based on data regarding resource utilization of the Bright Bodies program and participants' use of relevant medical and non-medical resources.

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoosh (Mona) Sharifi, MD, MPH, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Maine Medical Center, Portland, Maine

IPD SHARING:
Plan to Share IPD: No